CLINICAL TRIAL: NCT01504659
Title: Intranasal Ketamine In the Treatment of Pediatric Bipolar Disorder
Acronym: IKBP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative issues
Sponsor: Juvenile Bipolar Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JBRF001
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; treatment resistance; depression; ketamine; intranasal; child
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bipolar-Ketalar (Active Comparator): Children with a diagnosis of BP-I, BP-II or BP-NOS will receive 4 administrations of intranasal ketalar
  Interventions: Drug: Ketamine hydrochloride injection
- Bipolar-Placebo (Placebo Comparator): Children with a diagnosis of BP-I, BP-II or BP-NOS will receive 4 administrations of placebo
  Interventions: Drug: Flat tonic water (e.g., Canada Dry Tonic Water)

INTERVENTIONS:
Drug: Ketamine hydrochloride injection — Separate dosing regimens will be applied depending on the weight of the child. Group A with minimum-maximum weight of 20 kg-40 kg will receive a fixed initial dose of 10 mg ketamine(0.25-0.5mg/kg)and will not exceed a maximum dose of 40 mg ketamine. Group B with minimum - maximum weight of 40.01kg-100kg will get a fixed initial dose of 20 mg ketamine(0.20-0.5mg/kg) and will not exceed a maximum dose of 120mg. ketamine. There will be 4 administrations of the drug at three day intervals. Titration upward will depend upon degree of side effects, improvement from baseline on primary measures, subjective opinion. Doses will be held constant as long as a therapuetic response, as measure of 80% improvement on YBOCS and YMRS, is reached.
  Other Names: Ketalar NDA 016812; Ketamine Hydrochloride Injection, Abbot Hospital, 074549; Ketamine Hdyrochloride Injection, Bioniche, 076092; Ketamine Hydrochloride Injection, Bedford, 074524; Calypsol; Ketalin; Ketamax; Ketanest; Ketava; Ketmin; Ketolar; Petar; Soon-Soon
  Arms: Bipolar-Ketalar
Drug: Flat tonic water (e.g., Canada Dry Tonic Water) — Separate dosing regimens will be applied depending on the weight of the child. Group A with minimum-maximum weight of 20 kg-40 kg will receive a fixed initial dose of 0.1cc placebo and not exceed a maximum dose of 0.4cc placebo. Group B with minimum - maximum weight of 40.01kg-100kg will get a fixed initial dose of 0.2cc placebo and will not exceed a maximum dose of 1.2cc. placebo. There will be 4 administrations of the placebo at three day intervals. Titration upward will depend upon degree of side effects, improvement from baseline on primary measures, and subjective opinion. Doses will be held constant as long as a therapuetic response, as a measure of 80% improvement on YBOCS and YMRS, is reached.
  Arms: Bipolar-Placebo

SUMMARY:
The investigators plan to evaluate the efficacy and safety of intranasal Ketalar (ketamine hydrochloride) in the treatment of primary symptom manifestations of pediatric bipolar disorder; Fear of Harm (FOH) phenotype. This phenotype represents those children who are most resistant to traditional treatments and suffer repeated hospitalizations. Primary symptoms include fearfulness, aggression secondary to threat, mood and/or arousal instability, and psychosis. In addition to evaluation of efficacy and safety, the investigators will also analyze whether therapeutic response depends upon the degree to which the subject fits the FOH phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 6-12;
2. DSM-IV bipolar disorder (BPI, BPII, BP-NOS, BP-FOH);
3. Treatment resistant - as defined by failure to adequately respond to at least 2 different classes of medications such as mood stabilizers and antipsychotic agent.

Exclusion Criteria:

1. Contraindication to the use of ketamine, including allergy and current use of medicine contraindicated with ketamine;
2. Endocrine or neurological illness;
3. Previous history of closed head injury, current head injury associated with possible intracranial hypertension, central nervous system masses, abnormalities, or hydrocephalus, ever had loss of consciousness;
4. Previous history of glaucoma or acute globe injury
5. Abnormal nasal physiology which would not allow for adequate medication delivery;
6. Any change in medication type or dose within the past 30 days;
7. Treatment with any MAOI's currently or within the past 3 months;
8. Has had a course of ECT within the past 3 months;
9. Has ever used PCP or ketamine;
10. Meets DSM-IV criteria for Mental Retardation;
11. Has ever had Repetitive Transcranial Magnetic Stimulation (rTMS), Vagal Nerve Stimulation (VNS) or Deep Brain Stimulation;
12. Is currently hospitalized;
13. Has known or suspected schizophrenia, even if currently stable or controlled with medications
14. Is acutely suicidal or homicidal (i.e., in imminent danger with plan, urges and intent to harm oneself or others) including any serious attempts/those requiring hospitalization in the past 12 months or at the PI's discretion;
15. The presence of any abnormal laboratory findings or serious medical disorder or condition including: clinically significant organ system dysfunction; significant endocrine disease, including diabetes mellitus; hypothyroidism; cardiovascular disease (myocardial ischemia, heart failure, arrhythmias); coagulopathy; significant anemia; significant acute infection; glaucoma; dehydration; epilepsy; any intra-abdominal or intrathoracic surgery or limb amputation within the prior 6 months; any diagnosed cardiac condition causing documented hemodynamic compromise or dysfunction of the SA or AV node; any diagnosed respiratory condition causing documented or clinically recognized hypoxia (e.g., chronic obstructive or restrictive pulmonary disease); body weight approximately < 80% or > 120% ideal body weight; or any medical condition known to interfere with cognitive performance; medication-related exclusions include narcotic therapy, chronic acetaminophen use, acute sedative hypnotic withdrawal, corticosteroid or spironolactone therapy, regularly dosed narcotics or any other sedative therapy or medication that interferes with SA or AV node function or could be considered contraindicated with the sedative properties of ketamine.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale | Change from baseline at 8 days
Young Mania Rating Scale | Change from baseline at 11 days
Young Mania Rating Scale | Change from baseline at 14 days
Young Mania Rating Scale | Change from baseline at 17 days
Overt Aggression Scale | Change from baseline at day 8
Overt Aggression Scale | Change from baseline at day 11
Overt Aggression Scale | Change from baseline at day 14
Overt Aggression Scale | Change from baseline at day 17
Yale Brown Obsessive Compulsive Scale | Change from baseline at Day 18, aggressive and obsessive questions

SECONDARY OUTCOMES:
Wechsler Intelligence Scale for Children-IV | Change from baseline at day 18
Peripheral Thermal Challenge | Change from baseline on days 6, 7, 15 and 16
body temperature | Change from baseline over 16 hours spanning days 6-7 and 15-16.
  A proprietary ambulatory monitor will measure skin and tympanic temperature using conventional thermistors and IR sensors
Triaxial acceleration | Change from baseline over 16 hours spanning days 6-7 and 15-16.
  A proprietary ambulatory monitor will measure triaxial acceleration from the forehead using a commercially-available sensor that also provides a plethysmograph signal from which heart rate can be derived.
SpO2 | Change from baseline over 16 hours spanning days 6-7 and 15-16.
  A proprietary ambulatory monitor will measure triaxial acceleration from the forehead using a commercially-available sensor that also provides a plethysmograph signal from which heart rate can be derived.
Galvanic skin response | Change from baseline over 16 hours spanning days 6-7 and 15-16.
  A proprietary ambulatory monitor will measure galvanic skin response obtained with two conventional electrodes.
Delis-Kaplin Executive Function System | Change from baseline on day 18
Conner's Continuous Performance Test | Change from baseline on day 18
SCARED | change from baseline at day 18

CONTACTS AND LOCATIONS:
Overall Officials: Demitri Papolos, MD, Principal Investigator — Juvenile Bipolar Research Foundation
Locations (4):
- United States (4):
  - Individual homes of subjects, Not Predetermined, Connecticut
  - Juvenile Bipolar Research Foundation, Maplewood, New Jersey
  - Individual homes of subjects, Not Predetermined, New Jersey
  - Individual homes of subjects, Not Predetermined, New York

REFERENCES:
- See also: Juvenile Bipolar Research Foundation — http://www.jbrf.org/
- See also: Fear of harm, a possible phenotype of pediatric bipolar disorder — http://www.jbrf.org/librarydocs/correctedproof-7-23-09.pdf
- See also: Diagnostic Assessment Program for Juvenile Bipolar Disorder — http://www.jbrf.org/cpp/index.html
- See also: A strategy for identifying phenotypic subtypes — http://www.jbrf.org/librarydocs/JADPhenotypeArticle.pdf